CLINICAL TRIAL: NCT01722487
Title: Randomized, Multicenter, Open-label, Phase 3 Study of the Bruton's Tyrosine Kinase Inhibitor Ibrutinib Versus Chlorambucil in Patients 65 Years or Older With Treatment-naive Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: Open-label Phase 3 BTK Inhibitor Ibrutinib vs Chlorambucil Patients 65 Years or Older With Treatment-naive CLL or SLL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1115-CA; 2012-003967-23 (EudraCT Number)
Record Dates: First submitted 2012-10-29; First posted 2012-11-06 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CLL, SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibrutinib (Experimental): Ibrutinib will be supplied as hard gelatin 140-mg capsules for oral (PO) administration. Ibrutinib 420 mg (3 x 140-mg capsules) is administered orally once daily. The first dose will be delivered in the clinic on Day 1, after which subsequent dosing is typically on an outpatient basis. Ibrutinib will be dispensed to patients in bottles at each visit.
  Interventions: Drug: Ibrutinib
- Chlorambucil (Active Comparator): Chlorambucil will be supplied as 2-mg tablets for PO administration. Chlorambucil is administered orally on Days 1 and 15 of each 28-day cycle.The starting dosage (Cycle 1) is 0.5 mg/kg. If well tolerated, the Chlorambucil dose can be increased starting at Cycle 2, with increments of 0.1 mg/kg on Day 1 of each cycle to a maximum of 0.8 mg/kg.
  Interventions: Drug: Chlorambucil

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be supplied as hard gelatin 140-mg capsules for oral (PO) administration. Ibrutinib 420 mg (3 x 140-mg capsules) is administered orally once daily. The first dose will be delivered in the clinic on Day 1, after which subsequent dosing is typically on an outpatient basis. Ibrutinib will be dispensed to patients in bottles at each visit.
  Arms: Ibrutinib
Drug: Chlorambucil — Chlorambucil will be supplied as 2-mg tablets for PO administration. Chlorambucil is administered orally on Days 1 and 15 of each 28-day cycle. The starting dosage (Cycle 1) is 0.5 mg/kg. If well tolerated, the Chlorambucil dose can be increased starting at Cycle 2, with increments of 0.1 mg/kg on Day 1 of each cycle to a maximum of 0.8 mg/kg.
  Arms: Chlorambucil

SUMMARY:
A Randomized, Multicenter, Open-label, Phase 3 Study of the Bruton's Tyrosine Kinase Inhibitor PCI-32765 versus Chlorambucil in Patients 65 Years or Older with Treatment-naive Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma.

DETAILED DESCRIPTION:
Study design: This is a randomized, multicenter, open-label, Phase 3 study designed to compare the safety and efficacy of Ibrutinib versus Chlorambucil in treatment-naive patients 65 years or older who have CLL or SLL.

Eligible patients will be randomized in a 1:1 ratio to Treatment Arm A or B:

* Treatment Arm A: Oral Chlorambucil 0.5 mg/kg on Days 1 and 15 of each 28-day cycle; the dose can be increased, if well tolerated, in increments of 0.1 mg/kg on Day 1 of each cycle to a maximum of 0.8 mg/kg; patients receive a minimum of 3 and a maximum of 12 cycles, in the absence of progressive disease or unacceptable toxicity.
* Treatment Arm B: Oral Ibrutinib 420 mg/day Randomization will be stratified on Eastern Cooperative Oncology Group (ECOG) performance status (0,1 versus 2); presence of advanced Rai stage (yes/no), advanced being defined as Stages 3-4; and geographic region: US versus non-US.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of 65 years of age or greater. Patients between the ages of 65 and 70 years of age must have 1 or more of the following comorbidities that may preclude the use of frontline chemo-immunotherapy with fludarabine, cyclophosphamide, or rituximab:

   * creatinine clearance < 70 mL/min using the Cockcroft-Gault equation
   * platelet count < 100,000/μL or hemoglobin < 10 g/dL
   * clinically apparent autoimmune cytopenia (autoimmune hemolytic anemia or immune thrombocytopenia)
   * ECOG performance score = 1 or 2
2. Diagnosis of CLL/SLL that meets IWCLL diagnostic criteria (Hallek 2008)
3. Active disease meeting at least 1 of the following IWCLL criteria (Hallek 2008) for requiring treatment:

   * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia Massive, progressive, or symptomatic splenomegaly
   * Massive nodes or progressive or symptomatic lymphadenopathy
   * Progressive lymphocytosis
   * Autoimmune hemolytic anemia and/or immune thrombocytopenia that is poorly responsive to corticosteroids or standard therapy
   * Constitutional symptoms
4. Measurable nodal disease by computed tomography (CT)
5. ECOG performance status of 0-2
6. Life expectancy > 4 months from randomization
7. Adequate hematologic function, defined as absolute neutrophil count (ANC) ≥ 1,000/μL (independent of growth factor support for at least 7 days prior to screening) and platelet count ≥ 50,000/μL (independent of transfusion and growth factor support for at least 7 days prior to screening)
8. Adequate hepatic function, defined as serum aspartate transaminase (AST) and alanine transaminase (ALT) < 2.5 x upper limit of normal (ULN), and total bilirubin ≤ 1.5 x ULN
9. Adequate renal function, defined as estimated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation
10. Willingness to receive all outpatient treatment, all laboratory monitoring, and all radiological evaluations at the institution that administers study drug for the entire study
11. Willingness of male patients, if sexually active with a female of childbearing potential, to use an effective barrier method of contraception during the study and for 3 months following the last dose of study drug
12. Ability to provide written informed consent and to understand and comply with the requirements of the study

Exclusion Criteria:

1. Known involvement of the central nervous system by lymphoma or leukemia
2. History or current evidence of Richter's transformation or prolymphocytic leukemia
3. Documentation of deletion of the short arm of chromosome 17: del(17p13.1) in more than 20% of cells examined on any pretreatment fluorescence in situ hybridization (FISH) or cytogenetic evaluation
4. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura
5. Any previous treatment (chemotherapy, radiotherapy, and/or monoclonal antibodies) intended specifically to treat CLL/SLL
6. Received any immunotherapy, vaccine, or investigational drug within 4 weeks prior to randomization
7. Corticosteroid use within 1 week prior to first dose of study drug, with the exception of inhaled, topical, or other local administrations. Patients requiring systemic steroids at daily doses > 20 mg prednisone (or corticosteroid equivalent, see Appendix N), or those who are administered steroids for leukemia control or white blood cell (WBC)-count-lowering are excluded.
8. Major surgery within 4 weeks prior to randomization
9. History of prior malignancy, with the exception of the following:

   * malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to screening and felt to be at low risk for recurrence by treating physician
   * adequately treated nonmelanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
   * adequately treated cervical carcinoma in situ without current evidence of disease
10. Currently active, clinically significant cardiovascular disease or a history of myocardial infarction within 6 months prior to randomization
11. Inability to swallow capsules or tablets, or disease significantly affecting gastrointestinal function
12. Uncontrolled active systemic fungal, bacterial, viral, or other infection or requirement for intravenous (IV) antibiotics
13. Known history of infection with human immunodeficiency virus (HIV)
14. Serologic status reflecting active hepatitis B or C infection
15. History of stroke or intracranial hemorrhage within 6 months prior to enrollment
16. Current life-threatening illness, medical condition, or organ-system dysfunction that could compromise patient safety or put the study at risk
17. Requirement for anticoagulation with warfarin
18. Requirement for treatment with a strong CYP3A4/5 and/or CYP2D6 inhibitor

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 269 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Styles, MD, Study Director — Pharmacyclics LLC.
Locations (108):
- United States (22):
  - Site Reference ID/Investigator #047, Duarte, California
  - Site Reference ID/Investigator #408, La Jolla, California
  - Site Reference ID/Investigator #720, Santa Rosa, California
  - Site Reference ID/Investigator #038, Stanford, California
  - Site Reference ID/Investigator #125, Atlanta, Georgia
  - Site Reference ID/Investigator #126, Chicago, Illinois
  - Site Reference ID/Investigator #071, Louisville, Kentucky
  - Site Reference ID/Investigator #307, Worcester, Massachusetts
  - Site Reference ID/Investigator #387, Ann Arbor, Michigan
  - Site Reference ID/Investigator #221, St Louis, Missouri
  - Site Reference ID/Investigator #712, Las Vegas, Nevada
  - Site Reference ID/Investigator #350, New Hyde Park, New York
  - Site Reference ID/Investigator #127, Rochester, New York
  - Site Reference ID/Investigator #656, Goldsboro, North Carolina
  - Site Reference ID/Investigator #734, Columbus, Ohio
  - Site Reference ID/Investigator #677, Portland, Oregon
  - Site Reference ID/Investigator #050, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator #032, Houston, Texas
  - Site Reference ID/Investigator #381, Laredo, Texas
  - Site Reference ID/Investigator #653, San Antonio, Texas
  - Site Reference ID/Investigator #404, Seattle, Washington
  - Site Reference ID/Investigator #731, Walla Walla, Washington
- Australia (10):
  - Site Reference ID/Investigator #654, Kogarah, New South Wales
  - Site Reference ID/Investigator #503, Woolloongabba, Queensland
  - Site Reference ID/Investigator #163, Bedford Park, South Australia
  - Site Reference ID/Investigator #555, Hobart, Tasmania
  - Site Reference ID/Investigator #193, Box Hill, Victoria
  - Site Reference ID/Investigator #556, Clayton, Victoria
  - Site Reference ID/Investigator #501, Fitzroy, Victoria
  - Site Reference ID/Investigator #715, Frankston, Victoria
  - Site Reference ID/Investigator #558, Geelong, Victoria
  - Site Reference ID/Investigator #170, Heidelberg, Victoria
- Belgium (7):
  - Site Reference ID/Investigator #164, Brussels, Brussells
  - Site Reference ID/Investigator #727, Yvoir, Namur
  - Site Reference ID/Investigator #560, Ghent, Oost-Vlaanderen
  - Site Reference ID/Investigator #559, Leuven, Vlaams Brabant
  - Site Reference ID/Investigator #628, Bruges, West-Vlaanderen
  - Site Reference ID/Investigator #561, Antwerp
  - Site Reference ID/Investigator #184, Brussells
- Canada (3):
  - Site Reference ID/Investigator #157, Calgary, Alberta
  - Site Reference ID/Investigator #018, Edmonton, Alberta
  - Site Reference ID/Investigator #159, Ottawa, Ontario
- China (5):
  - Site Reference ID/Investigator #674, Guangzhou, Guangdong
  - Site Reference ID/Investigator #671, Nanjing, Jiangsu
  - Site Reference ID/Investigator #675, Hangzhou, Zhejiang
  - Site Reference ID/Investigator #670, Beijing
  - Site Reference ID/Investigator #673, Beijing
- Czechia (3):
  - Site Reference ID/Investigator #564, Hradec Králové, Královéhradecký kraj
  - Site Reference ID/Investigator #562, Brno
  - Site Reference ID/Investigator #566, Plzen-Lochotin
- Ireland (3):
  - Site Reference ID/Investigator #572, Dublin
  - Site Reference ID/Investigator #570, Dublin
  - Site Reference ID/Investigator #571, Galway
- Israel (6):
  - Site Reference ID/Investigator #573, Haifa
  - Site Reference ID/Investigator #576, Haifa
  - Site Reference ID/Investigator #577, Jerusalem
  - Site Reference ID/Investigator #578, Nahariya
  - Site Reference ID/Investigator #575, Petah Tikva
  - Site Reference ID/Investigator #574, Ramat Gan
- Italy (9):
  - Site Reference ID/Investigator #583, Rome, Lazio
  - Site Reference ID/Investigator #522, Rozzano, Milano
  - Site Reference ID/Investigator #582, Novara, Piedmont
  - Site Reference ID/Investigator #527, Padua, Veneto
  - Site Reference ID/Investigator #580, Bologna
  - Site Reference ID/Investigator #584, Milan
  - Site Reference ID/Investigator #523, Milan
  - Site Reference ID/Investigator #581, Milan
  - Site Reference ID/Investigator #524, Modena
- New Zealand (5):
  - Site Reference ID/Investigator #589, Christchurch, Canterbury
  - Site Reference ID/Investigator #586, Hamilton, Waikato Region
  - Site Reference ID/Investigator #663, Auckland
  - Site Reference ID/Investigator #588, Auckland
  - Site Reference ID/Investigator #587, Wellington
- Poland (5):
  - Site Reference ID/Investigator #590, Lublin, Lublin Voivodeship
  - Site Reference ID/Investigator #592, Brzozowie, Podkarpackie Voivodeship
  - Site Reference ID/Investigator #591, Chorzów
  - Site Reference ID/Investigator #529, Gdansk
  - Site Reference ID/Investigator #531, Lodz
- Russia (2):
  - Site Reference ID/Investigator #707, Ryazan
  - Site Reference ID/Investigator #304, Yaroslavl
- Spain (6):
  - Site Reference ID/Investigator #536, Majadahonda, Madrid
  - Site Reference ID/Investigator #534, Barcelona
  - Site Reference ID/Investigator #533, Barcelona
  - Site Reference ID/Investigator #535, Barcelona
  - Site Reference ID/Investigator #604, Barcelona
  - Site Reference ID/Investigator #537, Madrid
- Turkey (Türkiye) (6):
  - Site Reference ID/Investigator #608, Ankara
  - Site Reference ID/Investigator #606, Ankara
  - Site Reference ID/Investigator #599, Istanbul
  - Site Reference ID/Investigator #714, Izmir
  - Site Reference ID/Investigator #601, Izmir
  - Site Reference ID/Investigator #602, Kayseri
- Ukraine (7):
  - Site Reference ID/Investigator #598, Simferopol, Autonomous Republic of Crimea
  - Site Reference ID/Investigator #597, Cherkasy, Cherkasy Oblast
  - Site Reference ID/Investigator #594, Dnipropetrovsk, Dnipropetrovsk Oblast
  - Site Reference ID/Investigator #725, Kharkiv, Kharkivs’ka Oblast’
  - Site Reference ID/Investigator #596, Lviv, Lviv Oblast
  - Site Reference ID/Investigator #595, Vinnytsia, Vinnytsia Oblast
  - Site Reference ID/Investigator #724, Zhytomyr, Zhytomyr Oblast
- United Kingdom (9):
  - Site Reference ID/Investigator #551, Bournemouth, Dorset
  - Site Reference ID/Investigator #544, London, England
  - Site Reference ID/Investigator #668, Oxford, England
  - Site Reference ID/Investigator #549, Colchester, Essex
  - Site Reference ID/Investigator #607, Cardiff, South Glamergon
  - Site Reference ID/Investigator #550, Leeds, Yorkshire
  - Site Reference ID/Investigator #721, Birmingham
  - Site Reference ID/Investigator #548, Nottingham
  - Site Reference ID/Investigator #367, Southampton

IPD SHARING:
Plan to Share IPD: No
We share this information with FDA and other authorities for the purposes of analyzing the study but not with other researchers

REFERENCES:
- [Derived] Abuhelwa AY, Almansour SA, Brown JR, Al-Shamsi HO, Abuhelwa Z, Kharaba Z, Bustanji Y, Semreen MH, Ali S, Alhuraiji A, McKinnon RA, Sorich MJ, Alzoubi KH, Hopkins AM. Statin use and survival in CLL/SLL treated with ibrutinib: pooled analysis of 4 randomized controlled trials. Blood Adv. 2025 Jul 22;9(14):3566-3575. doi: 10.1182/bloodadvances.2024015287. PMID 40266025
- [Derived] Barr PM, Owen C, Robak T, Tedeschi A, Bairey O, Burger JA, Hillmen P, Dearden C, Grosicki S, McCarthy H, Li JY, Offner F, Moreno C, Jermain M, Zhou C, Hsu E, Szoke A, Kipps TJ, Ghia P. Many People With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma Benefit From Ibrutinib Treatment Up To 8 Years: A Plain Language Summary. Future Oncol. 2023 Jan 9. doi: 10.2217/fon-2022-0898. Online ahead of print. PMID 36617990
- [Derived] Barr PM, Owen C, Robak T, Tedeschi A, Bairey O, Burger JA, Hillmen P, Coutre SE, Dearden C, Grosicki S, McCarthy H, Li JY, Offner F, Moreno C, Zhou C, Hsu E, Szoke A, Kipps TJ, Ghia P. Up to 8-year follow-up from RESONATE-2: first-line ibrutinib treatment for patients with chronic lymphocytic leukemia. Blood Adv. 2022 Jun 14;6(11):3440-3450. doi: 10.1182/bloodadvances.2021006434. PMID 35377947
- [Derived] Burger JA, Robak T, Demirkan F, Bairey O, Moreno C, Simpson D, Munir T, Stevens DA, Dai S, Cheung LWK, Kwei K, Lal I, Hsu E, Kipps TJ, Tedeschi A. Up to 6.5 years (median 4 years) of follow-up of first-line ibrutinib in patients with chronic lymphocytic leukemia/small lymphocytic lymphoma and high-risk genomic features: integrated analysis of two phase 3 studies. Leuk Lymphoma. 2022 Jun;63(6):1375-1386. doi: 10.1080/10428194.2021.2020779. Epub 2022 Jan 11. PMID 35014928
- [Derived] Allan JN, Shanafelt T, Wiestner A, Moreno C, O'Brien SM, Li J, Krigsfeld G, Dean JP, Ahn IE. Long-term efficacy of first-line ibrutinib treatment for chronic lymphocytic leukaemia in patients with TP53 aberrations: a pooled analysis from four clinical trials. Br J Haematol. 2022 Feb;196(4):947-953. doi: 10.1111/bjh.17984. Epub 2021 Dec 5. PMID 34865212
- [Derived] Coutre SE, Byrd JC, Hillmen P, Barrientos JC, Barr PM, Devereux S, Robak T, Kipps TJ, Schuh A, Moreno C, Furman RR, Burger JA, O'Dwyer M, Ghia P, Valentino R, Chang S, Dean JP, James DF, O'Brien SM. Long-term safety of single-agent ibrutinib in patients with chronic lymphocytic leukemia in 3 pivotal studies. Blood Adv. 2019 Jun 25;3(12):1799-1807. doi: 10.1182/bloodadvances.2018028761. PMID 31196847
- [Derived] Barr PM, Robak T, Owen C, Tedeschi A, Bairey O, Bartlett NL, Burger JA, Hillmen P, Coutre S, Devereux S, Grosicki S, McCarthy H, Li J, Simpson D, Offner F, Moreno C, Zhou C, Styles L, James D, Kipps TJ, Ghia P. Sustained efficacy and detailed clinical follow-up of first-line ibrutinib treatment in older patients with chronic lymphocytic leukemia: extended phase 3 results from RESONATE-2. Haematologica. 2018 Sep;103(9):1502-1510. doi: 10.3324/haematol.2018.192328. Epub 2018 Jun 7. PMID 29880603
- [Derived] Brown JR, Moslehi J, O'Brien S, Ghia P, Hillmen P, Cymbalista F, Shanafelt TD, Fraser G, Rule S, Kipps TJ, Coutre S, Dilhuydy MS, Cramer P, Tedeschi A, Jaeger U, Dreyling M, Byrd JC, Howes A, Todd M, Vermeulen J, James DF, Clow F, Styles L, Valentino R, Wildgust M, Mahler M, Burger JA. Characterization of atrial fibrillation adverse events reported in ibrutinib randomized controlled registration trials. Haematologica. 2017 Oct;102(10):1796-1805. doi: 10.3324/haematol.2017.171041. Epub 2017 Jul 27. PMID 28751558
- [Derived] Burger JA, Tedeschi A, Barr PM, Robak T, Owen C, Ghia P, Bairey O, Hillmen P, Bartlett NL, Li J, Simpson D, Grosicki S, Devereux S, McCarthy H, Coutre S, Quach H, Gaidano G, Maslyak Z, Stevens DA, Janssens A, Offner F, Mayer J, O'Dwyer M, Hellmann A, Schuh A, Siddiqi T, Polliack A, Tam CS, Suri D, Cheng M, Clow F, Styles L, James DF, Kipps TJ; RESONATE-2 Investigators. Ibrutinib as Initial Therapy for Patients with Chronic Lymphocytic Leukemia. N Engl J Med. 2015 Dec 17;373(25):2425-37. doi: 10.1056/NEJMoa1509388. Epub 2015 Dec 6. PMID 26639149
- See also: www.pharmacyclics.com — http://www.pharmacyclics.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib: Ibrutinib 420 mg daily.
- Chlorambucil: Chlorambucil 0.5 mg/kg (to maximum 0.8 mg/kg) days 1 and 15 of 28-day cycle up to 12 cycles
Period: Overall Study
Arm/Group | Ibrutinib | Chlorambucil
Started | 136 | 133
Completed | 134 (Participants who were still on study or died at study closure) | 126 (Participants who were still on study or died at study closure)
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrutinib | Chlorambucil | Total
Number analyzed (Participants) | 136 | 133 | 269
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 136 | 133 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (5.67) | 73.4 (5.95) | 73.3 (5.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 88 | 81 | 169

OUTCOME MEASURES:

1. Primary Outcome: PFS (Progression Free Survival)
Description: The primary objective of this study was to evaluate the efficacy of Ibrutinib compared with Chlorambucil based on the independent review committee (IRC) assessment of PFS
  Progressive disease according to 2008 IWCLL guidelines was defined as:
  * Group A
    * Lymphadenopathy, increase ≥50%
    * Hepatomegaly, increase ≥50%
    * Splenomegaly, increase ≥50%
    * Blood lymphocytes, increase ≥ 50% over baseline
  * Group B
    * Platelets counts, decrease of ≥ 50% from baseline secondary to CLL
    * Hemoglobin, decrease of > 2 g/dL from baseline secondary to CLL
Time Frame: Analysis was conducted when 15 months had elapsed after the last subject was randomized with the cutoff date of 4 May 2015. The median follow-up time is 18 month.
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
Months | NA [NA to NA] — IBR: Median PFS was not reached so 95% CI for median PFS is not applicable. | 18.9 [14.1 to 22.0]
Statistical Analysis 1: Comparison: Chlorambucil; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.16, 95% CI 2-sided [0.09 to 0.28]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is calculated for all randomized subjects as the duration of time from the date of randomization to the date of death due to any cause or the date last known alive for subjects who were not known to have died at study closure.
Time Frame: as for outcome 1
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
Months | NA [NA to NA] — IBR: Median OS was not reached so 95% CI for median OS is not applicable. | NA [NA to NA] — CHL: Median OS was not reached so 95% CI for median OS is not applicable.
Statistical Analysis 1: Comparison: Chlorambucil; Test type: Superiority or Other; p = 0.0010, Log Rank; Hazard Ratio (HR) = 0.16, 95% CI 2-sided [0.05 to 0.56]

3. Secondary Outcome: ORR (Overall Response Rate)
Description: ORR is defined as the proportion of subjects who achieved complete response (CR), complete response with incomplete marrow recovery (CRi), nodule partial response (nPR) or PR per IRC assessment. Response criteria are as outlined in the International Workshop on CLL (iwCLL) 2008 criteria with the 2012 iwCLL modification stating that treatment-related lymphocytosis in the setting of improvement in other parameters was not considered as PD and the 2013 iwCLL clarification of criteria for a partial response to therapy.
Time Frame: as for outcome 1
Population: Intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
percentage of participants | 82.4 | 35.3
Statistical Analysis 1: Comparison: Chlorambucil; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Proportion of Sustained Hemoglobin Improvement
Description: The proportion of subjects who achieved Hemoglobin >11 g/dL or increase ≥ 2 g/dL over baseline and persisted continuously for ≥56 days (8 weeks) without blood transfusion or growth factors.
Time Frame: as for outcome 1
Population: Intention to treat
Measure: Number; unit: Percentage of Participants
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
Percentage of Participants | 45.6 | 20.3
Statistical Analysis 1: Comparison: Chlorambucil; Test type: Superiority or Other; p < 0.0001, Chi-squared

5. Secondary Outcome: Proportion of Sustained Hemoglobin Improvement in Subjects With Baseline Anemia
Description: In randomized subjects with baseline hemoglobin ≤ 11 g/dL, the proportion of subjects who achieved Hemoglobin >11 g/dL or increase ≥ 2 g/dL over baseline persisted continuously for ≥56 days (8 weeks) without blood transfusion or growth factors.
Time Frame: as for outcome 1
Population: Subjects with Baseline Anemia
Measure: Number; unit: Percentage of Participants
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 51 | 55
Percentage of Participants | 84.3 | 45.5
Statistical Analysis 1: Comparison: Chlorambucil; Test type: Superiority or Other; p < 0.0001, Chi-squared

6. Secondary Outcome: Proportion of Sustained Platelet Improvement
Description: The proportion of subjects who achieved platelet >100 x 10^9/L or increase ≥50% over baseline and persisted continuously for ≥56 days (8 weeks) without blood transfusion or growth factors.
Time Frame: as for outcome 1
Population: Intention to treat
Measure: Number; unit: Percentage of Participants
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
Percentage of Participants | 27.2 | 11.3
Statistical Analysis 1: Comparison: Chlorambucil; Test type: Superiority or Other; p = .0009, Chi-squared

7. Secondary Outcome: Proportion of Sustained Platelet Improvement in Subjects With Baseline Thrombocytopenia
Description: In randomized subjects with baseline platelet ≤ 100 x 10^9/L, the proportion of subjects who achieved platelet >100 x 10^9/L or increase ≥50% over baseline persisted continuously for ≥56 days (8 wee without blood transfusion or growth factors.
Time Frame: Analysis was conducted when 15 months had elapsed after the last subject was randomized with cutoff date of 4 May 2015. The median follow-up time is 18 month.
Population: Subjects With Baseline Thrombocytopenia
Measure: Number; unit: Percentage of Participants
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 35 | 28
Percentage of Participants | 77.1 | 42.9
Statistical Analysis 1: Comparison: Chlorambucil; Test type: Superiority or Other; p = .0054, Chi-squared

ADVERSE EVENTS:
Time Frame: From first dose of study drug to within 30 days of last dose or starting new anti-cancer therapy, whichever occurs earlier, up to 04May2015 ( data cutoff date for final analysis).
Description: 269 subjects were randomized on the study of which 2 subjects withdrew without treatment and were not included in the number of participants at risk. Investigators assess the occurrence of AEs and SAEs at all patient evaluation time points during the study.
Groups:
- PCI-32765: Ibrutinib 420 mg daily.
Arm/Group | PCI-32765 | Chlorambucil
Serious Adverse Events (participants affected / at risk) | 55/135 | 33/132
Other Adverse Events (participants affected / at risk) | 133/135 | 123/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765 (N=135) | Chlorambucil (N=132)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 2 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Aortic valve disease mixed (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 2 | 0
Hyphaema (Eye disorders) | 1 | 0
Retinal vascular occlusion (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 5
Chills (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Immunodeficiency (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 2
Bronchopneumonia (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Abscess limb (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Acute hepatitis B (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Heart rate irregular (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 0
Somatoform disorder cardiovascular (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765 (N=135) | Chlorambucil (N=132)
Anaemia (Blood and lymphatic system disorders) | 24 | 27
Neutropenia (Blood and lymphatic system disorders) | 20 | 29
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 17
Increased tendency to bruise (Blood and lymphatic system disorders) | 8 | 4
Atrial fibrillation (Cardiac disorders) | 7 | 0
Dry eye (Eye disorders) | 23 | 6
Lacrimation increased (Eye disorders) | 18 | 8
Vision blurred (Eye disorders) | 18 | 10
Visual acuity reduced (Eye disorders) | 15 | 3
Eye pain (Eye disorders) | 8 | 2
Vitreous floaters (Eye disorders) | 8 | 6
Cataract (Eye disorders) | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 57 | 22
Nausea (Gastrointestinal disorders) | 30 | 52
Constipation (Gastrointestinal disorders) | 20 | 21
Vomiting (Gastrointestinal disorders) | 18 | 27
Abdominal pain (Gastrointestinal disorders) | 17 | 14
Dyspepsia (Gastrointestinal disorders) | 15 | 3
Stomatitis (Gastrointestinal disorders) | 11 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 1
Fatigue (General disorders) | 41 | 50
Oedema peripheral (General disorders) | 25 | 12
Pyrexia (General disorders) | 22 | 17
Asthenia (General disorders) | 10 | 5
Upper respiratory tract infection (Infections and infestations) | 22 | 23
Urinary tract infection (Infections and infestations) | 13 | 10
Conjunctivitis (Infections and infestations) | 11 | 3
Nasopharyngitis (Infections and infestations) | 10 | 6
Cellulitis (Infections and infestations) | 8 | 1
Sinusitis (Infections and infestations) | 7 | 1
Skin infection (Infections and infestations) | 7 | 3
Herpes zoster (Infections and infestations) | 0 | 7
Contusion (Injury, poisoning and procedural complications) | 11 | 2
Weight decreased (Investigations) | 14 | 16
Platelet count decreased (Investigations) | 7 | 6
Decreased appetite (Metabolism and nutrition disorders) | 13 | 19
Hyperuricaemia (Metabolism and nutrition disorders) | 8 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2
Headache (Nervous system disorders) | 16 | 13
Dizziness (Nervous system disorders) | 15 | 16
Insomnia (Psychiatric disorders) | 11 | 9
Anxiety (Psychiatric disorders) | 7 | 2
Haematuria (Renal and urinary disorders) | 8 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 13 | 5
Night sweats (Skin and subcutaneous tissue disorders) | 9 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 3
Hypertension (Vascular disorders) | 18 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No